CLINICAL TRIAL: NCT05869045
Title: The Impact of Point-of-care Ultrasound (POCUS) on the Prognosis of Respiratory Failure in Patients Presenting to the Emergency Department Based on Diaphragmatic Dysfunction
Brief Title: POCUS and Respiratory Failure Prognosis Based on Diaphragmatic Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Carmine Cristiano Di Gioia, Attending physician, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: DSF
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Failure; Diaphragm Disease
Keywords: Point of care ultrasound; Diaphragm Disease
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Diaphragmatic dysfunction (DD): Patients with diaphragmatic dysfunction measured by point-of-care ultrasound using the diaphragm shortening fraction (DSF) method, which resulted in values lower than 10%. DSF is calculated by the formula: diaphragmatic thickness at the end of inspiration - diaphragmatic thickness at the end of expiration/diaphragmatic thickness at the end of expiration×100
  Interventions: Other: Diaphragm shortening fraction measurement by point-of-care ultrasound.
- Patients without Diaphragmatic dysfunction (DD): Patients without diaphragmatic dysfunction measured by point-of-care ultrasound using the DSF method, which resulted in values higher than 10%.
  Interventions: Other: Diaphragm shortening fraction measurement by point-of-care ultrasound.

INTERVENTIONS:
Other: Diaphragm shortening fraction measurement by point-of-care ultrasound. — A noninvasive and feasible method to assess diaphragmatic function and predict the prognosis of patients with respiratory failure presenting to the emergency department. The method consists of measuring the diaphragmatic thickness at the end of inspiration and expiration using a linear probe placed in the subcostal region and calculating the percentage of change using the formula: diaphragmatic thickness at the end of inspiration - diaphragmatic thickness at the end of expiration/diaphragmatic thickness at the end of expiration×100. A value lower than 10% indicates diaphragmatic dysfunction and a higher risk of adverse outcomes.

SUMMARY:
This study aims to evaluate the use of POCUS to assess diaphragmatic function and its association with clinical outcomes in patients with respiratory failure who are admitted to the emergency department.

DETAILED DESCRIPTION:
Respiratory failure is a common condition that requires prompt diagnosis and treatment in the emergency department. Diaphragmatic dysfunction (DD) is a potential contributor to respiratory failure, but it is often underdiagnosed and undertreated. Point-of-care ultrasound (POCUS) is a non-invasive and feasible tool that can measure diaphragmatic function using parameters such as diaphragm excursion and diaphragm shortening fraction (DSF). However, the prognostic value of POCUS for DD in patients with respiratory failure is unclear.

This study is a prospective observational cohort study that will enroll consecutive patients with respiratory failure who are admitted to the emergency department of a tertiary hospital. All patients will undergo POCUS examination of the diaphragm within 6 hours of admission by trained emergency physicians. The primary outcome will be the composite of mortality, intubation, or noninvasive ventilation failure within 30 days of admission. The secondary outcomes will include length of hospital stay, intensive care unit admission, and ventilator-free days. The association between POCUS parameters of diaphragmatic function and clinical outcomes will be analyzed using multivariate logistic regression and Cox proportional hazards models.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory failure defined as one or more of the following: respiratory rate >24 breaths/min, oxygen saturation <90% on room air, PaO2/FiO2 ratio <300 mmHg, or need for supplemental oxygen
* Ability to provide informed consent or availability of a legal representative

Exclusion Criteria:

* Pregnancy
* History of thoracic surgery or trauma
* Known neuromuscular disease affecting the diaphragm
* Contraindications for POCUS examination such as chest wall deformity, subcutaneous emphysema, or skin infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with respiratory failure who are admitted to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite of mortality, intubation, or noninvasive ventilation failure within 30 days of admission | Patients will be followed up for a maximum of 1 months from admission to the emergency department, until discharge or death

IPD SHARING:
Plan to Share IPD: Undecided